CLINICAL TRIAL: NCT04473456
Title: Combined Simultaneous EGD-colonoscopy (CoSi Endoscopy) Harmlessly Reduces Procedure Times: a Randomized Control Trial
Brief Title: Combined Simultaneous EGD-colonoscopy Trial (CoSi Endoscopy)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: EmuraCenter LatinoAmerica (Network)
Collaborators: Universidad de la Sabana (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: 2020-ECL-6-1
Record Dates: First submitted 2020-07-13; First posted 2020-07-16 (Actual); Last update posted 2020-12-08 (Actual); Status verified 2020-12

CONDITIONS: Procedure Time
Keywords: Combined simultaneous (CoSi) endoscopy; EGD; Colonoscopy
MeSH Terms: interventions — Colonoscopy

STUDY DESIGN:
Intervention Model Description: Patients are randomly assigned to non-intervention and intervention (simultaneous EGD and colonoscopy) arms
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Participants, care providers, and outcomes evaluator are masked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Serial arm (No Intervention): In the serial group, all colonoscopies will be performed by the same endoscopist. EGDs are performed by the attending endoscopist on the day of the procedure.
- Simultaneous arm (Active Comparator): In the simultaneous group, all colonoscopies will be performed by the same endoscopist. EGDs are performed by the attending endoscopist on the day of the procedure.
  Interventions: Procedure: Simultaneous EGD and colonoscopy

INTERVENTIONS:
Procedure: Simultaneous EGD and colonoscopy — Patients are examined simultaneously by EGD and colonoscopy
  Arms: Simultaneous arm

SUMMARY:
The COVID -19 pandemic has reduced endoscopy services to an average of 83% producing a significant economic impact on endoscopy units worldwide. Endoscopy as an aerosol-generating procedure requires endoscopy units to allow 12 cycles of air exchange per hour, equivalent to 20 minutes, between patients, to reduce medical risk exposure. Planning strategies to facilitate economic reactivation of endoscopy services in a responsible manner, maintaining adequate security measures for both patients and healthcare personnel is currently a major challenge. Serial endoscopic interventions as esophagogastroduodenoscopy (EGD) and colonoscopy are commonly performed during the same sedation time. Estimated times for quality inspection in the upper digestive tract and the colon, are 7 and 6 minutes, respectively. In addition, time to reach the cecum and to set up the following procedure increase not only procedure time but SARS-CoV-2 exposure to healthcare personnel. Performing these two procedures simultaneously by two endoscopists would considerably reduce procedure time while increasing the number of patients evaluated in one day, especially in the period of service reactivation. There are no studies comparing simultaneous EGD and colonoscopy procedures and, serial procedures. This study aims to determine differences in procedures times between simultaneous EGD-colonoscopy and conventional serial EGD-colonoscopy as an alternative to improve the number of procedures/hour/unit during the COVID-19 era.

DETAILED DESCRIPTION:
Study type:

This is a prospective controlled randomized study to determine differences in procedure times of simultaneous EGD-colonoscopy and serial EGD-colonoscopy. Patients are randomized into two groups: the serial group, where the EGD is performed first and thereafter the colonoscopy and, the simultaneous group, where the two procedures are performed at the same time, each by a trained gastroenterologist.

Patients:

Eligible patients are those consecutively scheduled for EGD and colonoscopy at EmuraCenter LatinoAmerica, Bogota DC, Colombia between June and August, 2020. Indications for procedures include among others abdominal pain, screening for digestive cancer, chronic anemia, digestive bleeding, and chronic diarrhea. Exclusion criteria are inadequate bowel preparation with Boston score with at least 1 point in any segment, residual gastric food, previous digestive system surgery, and refusal to participate. Patients and their accompanying person give written consent of the procedures and are asked to complete a telephone survey related to COVID-19 symptoms 1 day before the procedure and 30 minutes before the procedure.

Randomization:

Endoscopists participating in the study are experts endoscopists. In both groups, colonoscopies are performed by the same expert endoscopist. EGD in the serial group is performed by the attending endoscopist responsible for procedures that day.

Outcomes:

Variables to be compared between groups include unit entry's time, time to completion of both procedures, EGD time, EGD inspection time, colonoscopy time, time to teach the cecum, withdrawal time, inter-procedure time, unit's exit time, the dose of sedation agent and endoscopic findings. Oxygenation (pO2) and percutaneous pCo2 are evaluated 5 minutes before, 5, and 10 minutes during the procedure and 5 minutes after completing the last procedure. A trained physician or anesthesiologist will administrate sedation to patients using Propofol. Post-procedure symptoms will be assessed by written survey 30 minutes and 24 hours after the procedure. This survey evaluates 6 symptoms, 3 of which are related to sedation: Nausea, drowsiness, and dizziness. and, the other 3 symptoms are related to the endoscopic procedure: abdominal pain, bloating, and pharyngeal pain. Each of the 6 symptoms will be scored from 1 to 5 (1: None, 2: Mild, 3: Moderate, 4: Severe, and 5: Extreme).

Patient position and location of endoscopy systems:

All patients are positioned in the left lateral decubitus position. For simultaneous procedures, the EGD tower is located to the left side and the colonoscopy tower at the right side of the bedside at the level patient's head.

EGD:

The systematic complete photodocumentation approach proposed by Emura et al will be carried out to inspect the upper GI tract mucosa using a Fuji 7000 video processor and a Fuji Lasereo EG-760 gastroscope. BLI-bright digital chromoendoscopy will be performed to observe the hypopharynx, the esophagus, and the esophagogastric junction and, the LCI mode for evaluation of the stomach and duodenal mucosa. Low CO2 insufflation will be used using the Fuji GW-100 insufflator.

Colonoscopy in the serial group:

A Fuji Lasereo 7000 equipment and an EC-760ZP-V / L colonoscope will be used. The CO2 insufflation will be carried out with Fuji GW-100 equipment.

Colonoscopy in the parallel-group:

An Olympus Evis Exera II equipment and an H-180-AI colonoscope will be used. An Olympus UCR insufflator will be used for CO2 insufflation.

Transcutaneous measurement of pCo2:

The pCO2 measurements will be performed using a Tosca TCM kit (XLab Solutions). This equipment uses a transducer (ts sensor 54) that is positioned on the patient's arm and measures pCO2 non-invasively.

ELIGIBILITY:
Inclusion Criteria:

* Eligible patients are those scheduled for EGD and colonoscopy at EmuraCenter Latinoamerica, Bogota DC, Colombia between June and August 2020. Procedure indications: abdominal pain, chronic anemia, chronic diarrhea, cancer screening, gastrointestinal bleeding.

Exclusion Criteria:

* Exclusion criteria are inadequate bowel preparation with Boston score with at least 1 point in any segment, residual gastric food, previous surgery of the digestive tract, and refusal to participate.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2020-06-13 (Actual); Primary Completion 2020-09-22 (Actual); Study Completion 2020-09-23 (Actual)

PRIMARY OUTCOMES:
Procedures time | Time elapsed in minutes between the starting of the first procedure and the ending time of the second procedure in the serial arm or both procedures in the simultaneous arm.
  Time elapsed in minutes between the starting of the first procedure and the ending time of the second procedure in the serial arm or both procedures in the simultaneous arm.
Interprocedure time | Time elapsed in minutes between the end of the first procedure and the starting of the second procedure (only applies in serial arm)
  Time elapsed in minutes between the end of the first procedure and the starting of the second procedure (only applies in serial arm)
Upper GI inspection time | Time taken in minutes to inspect the entire upper GI mucosa according to the complete photodocumentation method proposed by Emura et al.
  Time taken in minutes to inspect the entire upper GI mucosa according to the complete photodocumentation method proposed by Emura et al.
Colonoscopy withdrawal time | Time elapsed in minutes between the cecum and the lower rectum used to inspect the colorectal mucosa
  Time elapsed in minutes between the cecum and the lower rectum used to inspect the colorectal mucosa
Colonoscopy insertion time | Time elapsed in minutes to reach the cecum
  Time elapsed in minutes to reach the cecum
EGD time | Time elapsed in minutes between the insertion of the gastroscope into the mouth and the extraction from the mouth
  Time elapsed in minutes between the insertion of the gastroscope into the mouth and the extraction from the mouth
Colonoscopy time | Time elapsed in minutes between the insertion of the colonoscope into the lower rectum and the extraction from the lower rectum
  Time elapsed in minutes between the insertion of the colonoscope into the lower rectum and the extraction from the lower rectum
Propofol used in EGD | Amount in mg of Propofol used during EGD
  Amount in mg of Propofol used during EGD
Propofol used in colonoscopy | Amount in mg of Propofol used during colonoscopy
  Amount in mg of Propofol used during colonoscopy
Propofol used in EGD and colonoscopy | Amount of Propofol in mg used fro procedures in the simultaneous arm
  Amount of Propofol in mg used fro procedures in the simultaneous arm.
percutaneous pCO2 | Measurement of pCO2 by the percutaneous transducer at 5 minutes prior and 5, 10 during procedures and 5 and 10 minutes minutes after completing the last procedure.
  Measurement of pCO2 by the percutaneous transducer at 5 minutes prior and 5, 10 during procedures and 5 and 10 minutes minutes after completing the last procedure.
percutaneous pO2 | Measurement of pO2 by the percutaneous transducer at 5 minutes prior and 5, 10 during procedures and 5 and 10 minutes minutes after completing the last procedure.
  Measurement of pO2 by the percutaneous transducer at 5 minutes prior and 5, 10 during procedures and 5 and 10 minutes minutes after completing the last procedure.
Position change 1 | During colonoscopy
  Change of patient's position during colonoscopy. Yes or No answer
Position change 2 | During olonoscopy
  If occurred, how many times the position changed. Numerical variable.
Post procedure symptoms survey related to colonoscopy | 20 minutes after the last procedure and after 24 hours
  Nausea, drowsiness, and dizziness are scored by patients using a scale from 1 to 5 (1: None, 2: Mild, 3: Moderate, 4: Severe, and 5: Extreme).
Post procedure symptoms survey related to sedation | 20 minutes after the last procedure and after 24 hours
  Abdominal pain, bloating, and pharyngeal pain are scored by patients using a scale from 1 to 5 (1: None, 2: Mild, 3: Moderate, 4: Severe, and 5: Extreme).

CONTACTS AND LOCATIONS:
Overall Officials: FABIAN EMURA, PhD, Principal Investigator — EmuraCenter LatinoAmerica
Locations (1):
- EmuraCenter LatinoAmerica, Bogota, Cundinamarca, Colombia

IPD SHARING:
Plan to Share IPD: Yes
There is s plan to share IPD with other researchers
Supporting Information: Study Protocol, SAP, ICF
Time Frame: December 1, 2020, for 1 month
Access Criteria: free access
URL: http://emuracenter.org

REFERENCES:
- [Background] Emura F, Sharma P, Arantes V, Cerisoli C, Parra-Blanco A, Sumiyama K, Araya R, Sobrino S, Chiu P, Matsuda K, Gonzalez R, Fujishiro M, Tajiri H. Principles and practice to facilitate complete photodocumentation of the upper gastrointestinal tract: World Endoscopy Organization position statement. Dig Endosc. 2020 Jan;32(2):168-179. doi: 10.1111/den.13530. Epub 2019 Nov 6. PMID 31529547
- [Background] Parasa S, Reddy N, Faigel DO, Repici A, Emura F, Sharma P. Global Impact of the COVID-19 Pandemic on Endoscopy: An International Survey of 252 Centers From 55 Countries. Gastroenterology. 2020 Oct;159(4):1579-1581.e5. doi: 10.1053/j.gastro.2020.06.009. Epub 2020 Jun 11. No abstract available. PMID 32534934
- [Background] Guda NM, Emura F, Reddy DN, Rey JF, Seo DW, Gyokeres T, Tajiri H, Faigel D. Recommendations for the Operation of Endoscopy Centers in the setting of the COVID-19 pandemic - World Endoscopy Organization guidance document. Dig Endosc. 2020 Sep;32(6):844-850. doi: 10.1111/den.13777. Epub 2020 Aug 12. PMID 32569438
- [Background] Bisschops R, Areia M, Coron E, Dobru D, Kaskas B, Kuvaev R, Pech O, Ragunath K, Weusten B, Familiari P, Domagk D, Valori R, Kaminski MF, Spada C, Bretthauer M, Bennett C, Senore C, Dinis-Ribeiro M, Rutter MD. Performance measures for upper gastrointestinal endoscopy: a European Society of Gastrointestinal Endoscopy (ESGE) Quality Improvement Initiative. Endoscopy. 2016 Sep;48(9):843-64. doi: 10.1055/s-0042-113128. Epub 2016 Aug 22. No abstract available. PMID 27548885
- [Background] Trencheva K, Dhar P, Sonoda T, Lee S, Samuels J, Stein B, Milsom J. Physiologic effects of simultaneous carbon dioxide insufflation by laparoscopy and colonoscopy: prospective evaluation. Surg Endosc. 2011 Oct;25(10):3279-85. doi: 10.1007/s00464-011-1705-2. Epub 2011 May 24. PMID 21607827